CLINICAL TRIAL: NCT01696279
Title: A 3-part Open-label Study to Assess the Pharmacokinetics of Lanthanum Carbonate, Compare the Efficacy, Safety and Tolerability of 8 Weeks of Treatment With Lanthanum Carbonate and Calcium Carbonate Using a Crossover Design and Investigate the Efficacy and Safety of 8 Months of Treatment With Lanthanum Carbonate in Hyperphosphataemic Children and Adolescents Aged 10 Years to <18 Years With Chronic Kidney Disease on Dialysis
Brief Title: A Study to Assess the Pharmacokinetics of Lanthanum Carbonate, Investigate and Compare the Efficacy, Safety and Tolerability of Lanthanum Carbonate With Calcium Carbonate in Hyperphosphataemic Children and Adolescents With Chronic Kidney Disease on Dialysis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SPD405-207; 2012-000171-17 (EudraCT Number)
Record Dates: First submitted 2012-09-26; First posted 2012-10-01 (Estimated); Results first posted 2020-01-02 (Actual); Last update posted 2021-06-10 (Actual); Status verified 2021-05

CONDITIONS: Chronic Kidney Disease; Hyperphosphatemia
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hyperphosphatemia | interventions — lanthanum carbonate; Calcium Carbonate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lanthanum Carbonate (Experimental): Participants will receive lanthanum carbonate orally at a total daily dose of 1500 mg to 3000 mg divided and mixed equally between in three meals.
  Interventions: Drug: Lanthanum Carbonate
- Calcium Carbonate (Active Comparator): Participants will receive calcium carbonate orally at a total daily dose adjusted as appropriate, until the target serum phosphorus level is achieved or until a maximum daily dose of 6500 mg is reached.
  Interventions: Drug: Calcium Carbonate

INTERVENTIONS:
Drug: Lanthanum Carbonate — Lanthanum Carbonate 1500 mg to 3000 mg powder will be administered orally.
  Other Names: SPD405
  Arms: Lanthanum Carbonate
Drug: Calcium Carbonate — Calcium carbonate will be administered orally at a total daily dose based on standard clinical practice. The total daily dose may be adjusted as appropriate, until the target serum phosphorus level is achieved or until a maximum daily dose of 6500 mg is reached.
  Arms: Calcium Carbonate

SUMMARY:
The purpose of this study is to summarize the percentage of participants achieving age-specific Kidney Disease Outcomes Quality Initiative (KDOQI) targets for serum phosphorus in hyperphosphatemic children and adolescents with chronic kidney disease (CKD) who are on dialysis, following 8 weeks of treatment with lanthanum carbonate.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 10 years to less than (<) 18 years of age at the time of consent.
2. Participant or parent/legally authorized representative (LAR) understand and are able, willing, and likely to fully comply with the study procedures and restrictions defined in this protocol.
3. Male, or non-pregnant, non-lactating female who agrees to comply with any applicable contraceptive requirements of the protocol.
4. Established chronic kidney disease (CKD), on dialysis, and requires treatment for hyperphosphatemia with a phosphate binder.
5. Serum phosphorus levels after a washout period of up to 3 weeks as follows: Age <12 years: Serum phosphorus greater than (>) 6.0 mg/dL (1.94 mmol/L); Age 12 years and older: Serum phosphorus >5.5mg/dL (1.78mmol/L).
6. Ability to provide written, signed and dated (personally or via an LAR) informed consent/and assent, as applicable, to participate in the study.

Exclusion Criteria:

1. Current or recurrent disease (example [eg], cardiovascular, liver, unstable and uncontrolled gastrointestinal, malignancy, or other conditions) other than CKD or end-stage renal disease that could affect the action, absorption or disposition of the investigational product, or clinical or laboratory assessments.
2. Current or relevant history of physical or psychiatric illness, any medical disorder (except for CKD or end-stage renal disease and related co-morbidities) that may require treatment or make the participant unlikely to fully complete the study, or any condition that presents undue risk from the investigational product or procedures.
3. Unable to eat semi-solid foods or on Total Enteral Alimentation.
4. Known or suspected intolerance or hypersensitivity to the investigational product(s), closely related compounds, or any of the stated ingredients.
5. History of alcohol or other substance abuse within the last year.
6. Current use of any medication (including over-the-counter, herbal, or homeopathic preparations) that could affect (improve or worsen) the condition being studied, or could affect the action, absorption, or disposition of the investigational product(s), or clinical or laboratory assessment.
7. Weight and age of participant are outside of local applicable criteria for blood sample volume limits.
8. Use of another investigational product within 30 days prior to receiving the first dose of investigational product.

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 63 (Actual)
Dates: Start 2013-02-15 (Actual); Primary Completion 2018-11-16 (Actual); Study Completion 2018-11-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (22):
- Centro Infantil Del Rinon S.R.L, San Miguel de Tucumán, Tucumán Province, Argentina
- Chile (2):
  - Hospital Luis Calvo Mackenna, Santiago
  - Hospital Dr. Sotero del Rio, Santiago
- Czechia (2):
  - Fakultni nemocnice Ostrava, Ostrava
  - University Hospital Motol, Prague
- Germany (2):
  - Kinder-und Jugendklinik Erlangen, Erlangen
  - Medizinische Hochschule Hannover, Hanover
- Hungary (3):
  - Semmelweis Egyetem Altalanos Orvostudomanyi Kar, Budapest, Bokay Janos
  - Debreceni Egyetem Orvos- es Egeszsegtudomanyi Centrum, Debrecen
  - Szegedi Tudomanyegyetem Altalanos Orvostudomanyi Kar, Szeged
- Poland (4):
  - Uniwersytecki Dzieciecy Szpital Kliniczny, Bialystok
  - Uniwersytecki Szpital Dzieciecy w Krakowie, Klinika Nefrologii Dzieciecej ze Stacja Dializ, Krakow
  - NZOZ tri-Medica, Lodz
  - Uniwersytecki Szpital Kliniczny, Wroclaw
- Romania (2):
  - Spitalul Clinic de Urgenta pentru Copii Sf. Maria, Iași
  - Spitalul Clinic de Urgenta pentru Copii - Louis Turcanu, Timișoara
- Russia (3):
  - Children City Clinical Hospital of Saint Vladimir, Moscow
  - Saint-Petersburg State Budgetary Healthcare Institution "Children City Hospital #1", Saint Petersburg
  - State Budgetary Healthcare Instit. of Sverdiov Region "Regional Children Clinical Hosp #1", Yekaterinburg
- Turkey (Türkiye) (3):
  - Cukurova University Faculty of Medicine Paediatric Nephrology, Adana
  - Izmir Tepecik Training and Research Hospital, Izmir
  - Manisa Celal Bayar University Hafsa Sultan Hospital, Manisa

REFERENCES:
- [Derived] Wasilewska A, Murray RA, Sundberg A, Uddin S, Achenbach H, Shavkin A, Szabo T, Vergani A, Umeh O. An open-label phase 2 trial to assess the efficacy, safety and pharmacokinetics of lanthanum carbonate in hyperphosphatemic children and adolescents with chronic kidney disease undergoing dialysis. BMC Nephrol. 2022 Mar 2;23(1):84. doi: 10.1186/s12882-022-02688-9. PMID 35236302

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 23 study centers between 15 February 2013 (first participant first visit) and 16 November 2018 (last participant last visit).
Pre-assignment Details: It was a 3 part study (Part 1: Pharmacokinetic assessment, Part 2: [Part 2a-calcium carbonate and lanthanum carbonate {crossover comparison} or Part 2b-lanthanum carbonate], Part 3: lanthanum carbonate treatment for 6 months). Overall 63 participants enrolled in the study.
Groups:
- Part 1: Single Dose Lanthanum Carbonate: Participants aged 10 to 12 years received 500 milligram (mg) and greater than (>) 12 years received 1000 mg single dose of lanthanum carbonate oral powder in the morning following breakfast.
- Part 2a: Calcium Carbonate, Then Lanthanum Carbonate (8 Weeks): Participants received calcium carbonate oral tablet until the target serum phosphorus level achieved or until a maximum daily dose of 6500 mg was reached and once serum phosphorus control was achieved the dose was maintained until the end of 8 weeks calcium carbonate, followed by 3 weeks of washout period (if necessary). At the end of first 8-week treatment period of part 2a, participants received lanthanum carbonate powder orally at a daily dose of 1500 mg mixed into meals and given three times a day or twice daily with a single dose not exceeding 1000 mg, total daily dose was titrated bi-weekly until a maximum dose of 3000 mg was reached and once the serum phosphorus control was achieved the dose was maintained until the end of 8 weeks lanthanum carbonate treatment period.
- Part 2b: Lanthanum Carbonate (8 Weeks): Participants received lanthanum carbonate powder orally at a daily dose of 1500 mg mixed into meals and given three times a day or twice daily with a single dose not exceeding 1000 mg, total daily dose was titrated bi-weekly until a maximum dose of 3000 mg was reached and once the serum phosphorus control was achieved the dose was maintained until the end of 8 weeks (Part 2b).
- Part 3: Lanthanum Carbonate (6 Months): Participants who completed in Part 2 (2a or 2b) could continue to receive lanthanum carbonate for an additional 6 months. Dosage of lanthanum carbonate was determined by the investigator based on serum phosphate levels taken at each study visit up to a maximum dose of 3000 mg/day.
Period: Part 1: Single Dose Lanthanum Carbonate
Arm/Group | Part 1: Single Dose Lanthanum Carbonate | Part 2a: Calcium Carbonate, Then Lanthanum Carbonate (8 Weeks) | Part 2b: Lanthanum Carbonate (8 Weeks) | Part 3: Lanthanum Carbonate (6 Months)
Started | 20 | 0 | 0 | 0
Safety Analysis Set 1 | 20 | 0 | 0 | 0
Entered Part 2a | 19 | 0 | 0 | 0
Completed | 19 | 0 | 0 | 0
Not Completed | 1 | 0 | 0 | 0
Not completed — Kidney Transplant | 1 | 0 | 0 | 0
Period: Part 2a: Calcium Carbonate + Lanthanum
Arm/Group | Part 1: Single Dose Lanthanum Carbonate | Part 2a: Calcium Carbonate, Then Lanthanum Carbonate (8 Weeks) | Part 2b: Lanthanum Carbonate (8 Weeks) | Part 3: Lanthanum Carbonate (6 Months)
Started | 0 | 53 (19 participants enrolled from Part 1 and 34 new participants enrolled in Part 2a) | 0 | 0
Safety Completer Set | 0 | 37 | 0 | 0
Full Analysis Set | 0 | 53 | 0 | 0
Per-protocol Set 1 | 0 | 17 | 0 | 0
Per-protocol Set 2 | 0 | 25 | 0 | 0
Entered Part 3 | 0 | 34 | 0 | 0
Completed | 0 | 34 | 0 | 0
Not Completed | 0 | 19 | 0 | 0
Not completed — Adverse Event | 0 | 5 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0
Not completed — Protocol Violation | 0 | 1 | 0 | 0
Not completed — Other (Unspecified) | 0 | 3 | 0 | 0
Not completed — Kidney Transplant | 0 | 7 | 0 | 0
Not completed — Non-Compliance with Study Drug | 0 | 2 | 0 | 0
Period: Part 2b: Lanthanum Carbonate (8 Weeks)
Arm/Group | Part 1: Single Dose Lanthanum Carbonate | Part 2a: Calcium Carbonate, Then Lanthanum Carbonate (8 Weeks) | Part 2b: Lanthanum Carbonate (8 Weeks) | Part 3: Lanthanum Carbonate (6 Months)
Started | 0 | 0 | 9 (9 new participants were enrolled in Part 2b) | 0
Safety Completer Set | 0 | 0 | 9 | 0
Full Analysis Set | 0 | 0 | 9 | 0
Per-protocol Set 1 | 0 | 0 | 0 | 0
Per-protocol Set 2 | 0 | 0 | 9 | 0
Completed | 0 | 0 | 8 | 0
Not Completed | 0 | 0 | 1 | 0
Not completed — Kidney Transplant | 0 | 0 | 1 | 0
Period: Part 3: Lanthanum Carbonate (6 Months)
Arm/Group | Part 1: Single Dose Lanthanum Carbonate | Part 2a: Calcium Carbonate, Then Lanthanum Carbonate (8 Weeks) | Part 2b: Lanthanum Carbonate (8 Weeks) | Part 3: Lanthanum Carbonate (6 Months)
Started | 0 | 0 | 0 | 42 (34 participants from Part 2a and 8 participants from Part 2b continued to Part 3)
Completed | 0 | 0 | 0 | 34
Not Completed | 0 | 0 | 0 | 8
Not completed — Kidney transplant | 0 | 0 | 0 | 6
Not completed — Other (Unspecified) | 0 | 0 | 0 | 1
Not completed — Missing | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety analysis set 1 and 2 included all participants who had taken 1 dose of IP in Part 1 for SAS 1, Part 2 or 3 for SAS 2 and who had completed at least 1 follow-up safety assessment. Few participants were analyzed in multiple arms/periods within the study, hence to avoid the duplication, baseline was analyzed only for the overall participants.
Groups:
- Overall Study: Study was conducted in 3 parts, participants aged 10 to 12 years received 500 milligram (mg) and greater than (>) 12 years received 1000 mg single dose of lanthanum carbonate oral powder respectively during part 1, followed by part 2 during which participants received calcium carbonate tablet for 8 weeks until a maximum daily dose of 6500 mg was reached (part 2a-Treatment period 1) and then received lanthanum carbonate oral powder for 8 weeks until a daily dose of 1500 mg was reached (part 2a-Treatment period 2). Eligible participants received lanthanum carbonate oral powder for 8 weeks at a daily dose of 1500 mg, which was titrated bi-weekly until a daily dose of 3000 mg was achieved (part 2b). Participants who completed part 2 continued the same treatment for additional 6 months during the part 3.
Arm/Group | Overall Study
Number analyzed (Participants) | 63
Age, Continuous [Mean (Standard Deviation); unit: Year] | 13.1 (2.65)
Age, Customized [Count of Participants; unit: Participants]
  Age group: < 10 years | 3
  Age group: ≥10 to <12 years | 11
  Age group: ≥12 to <18 years | 49
  Age group: ≥18 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 36
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 58
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 61
  Black or African American | 0
  Native Hawaiian or other Pacific Islander | 0
  Asian | 0
  American Indian or Alaska Native | 0
  Multiple | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Age-Specific Kidney Disease Outcomes Quality Initiative (KDOQI) Targets for Serum Phosphate Level Following 8 Weeks of Lanthanum Carbonate Administration (Part 2 + Part 3)
Description: KDOQI serum phosphorus targets were defined for: Adolescents aged greater than or equal to (>=) 12 to less than (<) 18 years to be less than or equal to (<=) 5.5 milligrams per deciliter (mg/dL) (1.78 millimoles per liter [mmol/L]); Children aged >=10 years to <12 years to be <= 6.0 mg/dL (1.94 mmol/L). Percentage of participants achieving age-specific KDOQI targets for serum phosphate level was reported only for the participants who had received lanthanum carbonate during part 2 or part 3. Data was analyzed and presented as per the intervention received in this study related to this outcome and not analyzed based on each part of the study.
Time Frame: After 8 weeks of lanthanum carbonate administration in Part 2 and/or in Part 3
Population: Per-protocol set 2 (PP2) included participants who had taken at least 1 dose of investigational product and completed 8 weeks of treatment with lanthanum carbonate and who had serum phosphate assessment data available during Part 2 or Part 3 to allow summarizing the percentage of participants achieving age-specific KDOQI target.
Measure: Number; unit: Percentage of participants
Groups:
- Part 2 + Part 3: Lanthanum Carbonate: Participants received lanthanum carbonate powder at a daily dose of 1500 mg mixed into meals and given three times a day or twice daily with a single dose not exceeding 1000 mg, total daily dose was titrated bi-weekly until a maximum dose of 3000 mg was reached and once the serum phosphorus control was achieved the dose was maintained until the end of 8 weeks treatment period (Part 2a and Part 2b) and continued to receive lanthanum carbonate for additional 6 months (Part 3).
Arm/Group | Part 2 + Part 3: Lanthanum Carbonate
Number analyzed (Participants) | 34
Percentage of participants | 50

2. Secondary Outcome: Percentage of Participants Achieving Age-Specific Kidney Disease Outcomes Quality Initiative (KDOQI) Targets for Serum Phosphate Level During Part 2
Description: KDOQI serum phosphorus targets was defined for: Adolescents aged >= 12 < 18 years to be <= 5.5 mg/dL (1.78 [mmol/L]); Children aged >=10 years to <12 years to be <= 6.0 mg/dL (1.94 mmol/L). Percentage of participants achieving age-specific KDOQI targets for serum phosphate level were reported only for the participants who had received calcium carbonate followed by 8 weeks of treatment with lanthanum carbonate in Part 2. Data was analyzed and presented as per the intervention received in this study related to this outcome and not analyzed based on each part of the study.
Time Frame: Up to 19 weeks
Population: Per Protocol Set 1 (PP1) included participants who had taken at least 1 dose of investigational product and completed 8 weeks of calcium carbonate followed by 8 weeks of lanthanum carbonate and who had serum phosphate assessment data available during Part 2 to allow summarizing the percentage of participants achieving age-specific KDOQI target.
Measure: Number; unit: Percentage of participants
Groups:
- Part 2: Calcium Carbonate: Participants received calcium carbonate oral tablet until the target serum phosphorus level achieved or until a maximum daily dose of 6500 mg was reached and once serum phosphorus control was achieved the dose was maintained until the end of 8 weeks (Part 2a: treatment period 1).
- Part 2: Lanthanum Carbonate: Participants received lanthanum carbonate powder orally at a daily dose of 1500 mg mixed into meals and given three times a day or twice daily with a single dose not exceeding 1000 mg, once the serum phosphorus control was achieved the dose was maintained until the end of 8 weeks (Part 2a: treatment period 2), also participants received lanthanum carbonate powder orally at a daily dose of 1500 mg mixed into meals and given three times a day or twice daily with a single dose not exceeding 1000 mg, total daily dose was titrated bi-weekly until a maximum dose of 3000 mg was reached and once the serum phosphorus control was achieved the dose was maintained until the end of 8 weeks (Part 2b).
Arm/Group | Part 2: Calcium Carbonate | Part 2: Lanthanum Carbonate
Number analyzed (Participants) | 17 | 17
Percentage of participants | 58.8 | 70.6

3. Secondary Outcome: Change From Baseline in Serum Phosphorus Levels Following Treatment With Lanthanum Carbonate After 8 Weeks
Description: Changes from baseline in serum phosphorus levels in hyperphosphatemic children and adolescents with chronic kidney disease (CKD) who are on dialysis, following treatment with lanthanum carbonate for 8 weeks were combined and reported. Baseline was defined as the last assessment prior to the first dose of investigational product. Data was analyzed and presented as per the intervention received in this study related to this outcome and not analyzed based on each part of the study.
Time Frame: Baseline, Week 8 of lanthanum carbonate administration in Part 2 and/or in Part 3
Population: PP2 included participants who had taken at least 1 dose of investigational product and completed 8 weeks of treatment with lanthanum carbonate and who had serum phosphate assessment data available during Part 2 or Part 3 to allow summarizing the percentage of participants achieving age-specific KDOQI target.
Measure: Mean (Standard Error); unit: millimoles per liter (mmol/L)
Arm/Group | Part 2 + Part 3: Lanthanum Carbonate
Number analyzed (Participants) | 34
millimoles per liter (mmol/L) | -0.334 (0.1035)

4. Secondary Outcome: Change From Baseline in Calcium Levels Following Treatment With Lanthanum Carbonate After Week 8
Description: Changes from baseline in calcium levels in hyperphosphatemic children and adolescents with CKD who are on dialysis, following treatment with lanthanum carbonate for 8 weeks were combined and reported. Baseline was defined as the last assessment prior to the first dose of investigational product. Data was analyzed and presented as per the intervention received in this study related to this outcome and not analyzed based on each part of the study.
Time Frame: Baseline, Week 8 of lanthanum carbonate administration in Part 2 and/or in Part 3
Population: as for outcome 3
Measure: Mean (Standard Error); unit: millimole per liter (mmol/L)
Arm/Group | Part 2 + Part 3: Lanthanum Carbonate
Number analyzed (Participants) | 34
millimole per liter (mmol/L) | -0.001 (0.0363)

5. Secondary Outcome: Change From Baseline in Calcium-Phosphorus Product Levels Following Treatment With Lanthanum Carbonate After Week 8
Description: Changes from baseline in calcium-phosphorus product levels in hyperphosphatemic children and adolescents with CKD who are on dialysis, following treatment with lanthanum carbonate for 8 weeks were combined and reported. Baseline was defined as the last assessment prior to the first dose of investigational product. The unit of measure for this outcome measure was millimole square per square liter (mmol^2/L^2). Data was analyzed and presented as per the intervention received in this study related to this outcome and not analyzed based on each part of the study.
Time Frame: Baseline, Week 8 of lanthanum carbonate administration in Part 2 and/or in Part 3
Population: as for outcome 3
Measure: Mean (Standard Error); unit: mmol^2/L^2
Arm/Group | Part 2 + Part 3: Lanthanum Carbonate
Number analyzed (Participants) | 34
mmol^2/L^2 | -0.577 (0.2464)

6. Secondary Outcome: Change From Baseline in Serum Phosphorus Levels Following Treatment With Calcium Carbonate After 8 Weeks and Lanthanum Carbonate After 8 Weeks During Part 2
Description: Changes from baseline in serum phosphorus levels in hyperphosphatemic children and adolescents with CKD who are on dialysis, following treatment with calcium carbonate after 8 weeks and lanthanum carbonate after 8 weeks were combined and reported. Baseline was defined as the last assessment prior to the first dose of investigational product. Here, number of participants analyzed refers to the number of participants evaluable for this outcome at specified time point. Data was analyzed and presented as per the intervention received in this study related to this outcome and not analyzed based on each part of the study.
Time Frame: Baseline, Week 8
Population: PP1 included participants who had taken at least 1 dose of investigational product and completed 8 weeks of calcium carbonate followed by 8 weeks of lanthanum carbonate and who had serum phosphate assessment data available during Part 2 to allow summarizing the percentage of participants achieving age-specific KDOQI target.
Measure: Mean (Standard Error); unit: millimole per liter (mmol/L)
Arm/Group | Part 2: Calcium Carbonate | Part 2: Lanthanum Carbonate
Number analyzed (Participants) | 16 | 17
millimole per liter (mmol/L) | -0.520 (0.1786) | -0.467 (0.1312)

7. Secondary Outcome: Change From Baseline in Calcium Levels Following Treatment With Calcium Carbonate After 8 Weeks and Lanthanum Carbonate After 8 Weeks During Part 2
Description: Changes from baseline in calcium levels in hyperphosphatemic children and adolescents with CKD who are on dialysis, following treatment with calcium carbonate after 8 weeks and lanthanum carbonate after 8 weeks were combined and reported. Baseline was defined as the last assessment prior to the first dose of investigational product. Here, number of participants analyzed refers to the number of participants evaluable for this outcome at specified time point. Data was analyzed and presented as per the intervention received in this study related to this outcome and not analyzed based on each part of the study.
Time Frame: Baseline, Week 8
Population: as for outcome 6
Measure: Mean (Standard Error); unit: millimole per liter (mmol/L)
Arm/Group | Part 2: Calcium Carbonate | Part 2: Lanthanum Carbonate
Number analyzed (Participants) | 16 | 17
millimole per liter (mmol/L) | 0.058 (0.0554) | -0.009 (0.0574)

8. Secondary Outcome: Change From Baseline in Calcium-Phosphorus Product Levels Following Treatment With Calcium Carbonate After 8 Weeks and Lanthanum Carbonate After 8 Weeks During Part 2
Description: Changes from baseline in calcium-phosphorus product levels in hyperphosphatemic children and adolescents with CKD who are on dialysis, following treatment with calcium carbonate after 8 weeks and lanthanum carbonate after 8 weeks were combined and reported. Baseline was defined as the last assessment prior to the first dose of investigational product. The unit of measure for this outcome was millimole square per square liter. Here, number of participants analyzed refers to the number of participants evaluable for this outcome at specified time point. Data was analyzed and presented as per the intervention received in this study related to this outcome and not analyzed based on each part of the study.
Time Frame: Baseline, Week 8
Population: as for outcome 6
Measure: Mean (Standard Error); unit: mmol^2/L^2
Arm/Group | Part 2: Calcium Carbonate | Part 2: Lanthanum Carbonate
Number analyzed (Participants) | 16 | 17
mmol^2/L^2 | -0.966 (0.4084) | -0.669 (0.3834)

9. Secondary Outcome: Change From Baseline in Serum Phosphorus Levels at the Last Visit of 8-Week Treatment Period in Part 2 and Monthly During 6-Month Extension Phase of Part 3
Description: Change from baseline in serum phosphorus levels at the last visit of each 8-week treatment period during Part 2 and monthly during the 6-month extension phase (Part 3) were reported. Baseline was defined as the last assessment prior to the first dose of investigational product. Here, number of participants analyzed refers to the number of participants evaluable for this outcome at specified time point. Data was analyzed and presented as per the intervention received in this study related to this outcome and not analyzed based on each part of the study.
Time Frame: Baseline, Week 8, 12, 16, 20, 24, 28 and Week 32
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: millimole per liter (mmol/L)
Arm/Group | Part 2 + Part 3: Lanthanum Carbonate
Number analyzed (Participants) | 34
millimole per liter (mmol/L)
  Change at Week 8 | -0.334 (0.1035)
  Change at Week 12: number analyzed (Participants) | 30
  Change at Week 12 | -0.416 (0.0912)
  Change at Week 16: number analyzed (Participants) | 27
  Change at Week 16 | -0.314 (0.1278)
  Change at Week 20: number analyzed (Participants) | 25
  Change at Week 20 | -0.316 (0.1055)
  Change at Week 24: number analyzed (Participants) | 23
  Change at Week 24 | -0.322 (0.1356)
  Change at Week 28: number analyzed (Participants) | 20
  Change at Week 28 | -0.236 (0.1491)
  Change at Week 32: number analyzed (Participants) | 13
  Change at Week 32 | -0.143 (0.1558)

10. Secondary Outcome: Change From Baseline in Calcium Levels at the Last Visit of 8-Week Treatment Period in Part 2 and Monthly During 6-Month Extension Phase of Part 3
Description: Change from baseline in calcium levels at the last visit of each 8-week treatment period during Part 2 and monthly during the 6- month extension phase (Part 3) were reported.Baseline was defined as the last assessment prior to the first dose of investigational product. Here, number of participants analyzed refers to the number of participants evaluable for this outcome at specified time point. Data was analyzed and presented as per the intervention received in this study related to this outcome and not analyzed based on each part of the study.
Time Frame: Baseline, Week 8, 12, 16, 20, 24, 28 and Week 32
Population: as for outcome 3
Measure: Mean (Standard Error); unit: millimole per liter (mmol/L)
Arm/Group | Part 2 + Part 3: Lanthanum Carbonate
Number analyzed (Participants) | 34
millimole per liter (mmol/L)
  Change at Week 8 | -0.001 (0.0363)
  Change at Week 12: number analyzed (Participants) | 28
  Change at Week 12 | -0.045 (0.0475)
  Change at Week 16: number analyzed (Participants) | 26
  Change at Week 16 | -0.034 (0.0534)
  Change at Week 20: number analyzed (Participants) | 22
  Change at Week 20 | 0.003 (0.0511)
  Change at Week 24: number analyzed (Participants) | 22
  Change at Week 24 | -0.010 (0.0450)
  Change at Week 28: number analyzed (Participants) | 20
  Change at Week 28 | 0.049 (0.0623)
  Change at Week 32: number analyzed (Participants) | 13
  Change at Week 32 | -0.127 (0.0773)

11. Secondary Outcome: Change From Baseline in Calcium-Phosphorus Product Levels at the Last Visit of 8-Week Treatment Period in Part 2 and Monthly During 6-Month Extension Phase of Part 3
Description: Change from baseline in calcium-phosphorus product levels at the last visit of each 8-week treatment period during Part 2 and monthly during the 6-month extension phase (Part 3) were reported. Baseline was defined as the last assessment prior to the first dose of investigational product. Here, number of participants analyzed refers to the number of participants evaluable for this outcome at specified time point. The unit of measure of this outcome was millimole square per square liter. Data was analyzed and presented as per the intervention received in this study related to this outcome and not analyzed based on each part of the study.
Time Frame: Baseline, Week 8, 12, 16, 20, 24, 28 and Week 32
Population: as for outcome 3
Measure: Mean (Standard Error); unit: mmol^2/L^2
Arm/Group | Part 2 + Part 3: Lanthanum Carbonate
Number analyzed (Participants) | 34
mmol^2/L^2
  Change at Week 8 | -0.577 (0.2464)
  Change at Week 12: number analyzed (Participants) | 28
  Change at Week 12 | -0.783 (0.2535)
  Change at Week 16: number analyzed (Participants) | 26
  Change at Week 16 | -0.575 (0.3023)
  Change at Week 20: number analyzed (Participants) | 22
  Change at Week 20 | -0.362 (0.2711)
  Change at Week 24: number analyzed (Participants) | 22
  Change at Week 24 | -0.578 (0.3459)
  Change at Week 28: number analyzed (Participants) | 20
  Change at Week 28 | -0.326 (0.3767)
  Change at Week 32: number analyzed (Participants) | 13
  Change at Week 32 | -0.570 (0.3624)

12. Secondary Outcome: Change From Baseline in Biochemical Bone Markers
Description: Change from baseline in bone turnover markers including bone alkaline phosphatase (ALP), osteocalcin, and sclerostin was reported for combined Part 2 and 3. End of the study (EOS) was defined as the completion if the participants benefited from and desired to continue dosing with lanthanum. Here, number of participants analyzed refers to the number of participants evaluable for this outcome at specified time point. Data was analyzed and presented as per the intervention received in this study related to this outcome and not analyzed based on each part of the study.
Time Frame: Baseline, Week 8, Week 16 and EOS (up to 42 weeks)
Population: as for outcome 6
Measure: Mean (Standard Error); unit: microgram per liter (ug/L)
Arm/Group | Part 2: Calcium Carbonate | Part 2 + Part 3: Lanthanum Carbonate
Number analyzed (Participants) | 17 | 17
microgram per liter (ug/L)
  ALP : Change at Week 8: number analyzed (Participants) | 16 | 0
  ALP : Change at Week 8 | -0.78 (8.503) |
  ALP : Change at Week 16: number analyzed (Participants) | 0 | 15
  ALP : Change at Week 16 |  | 31.86 (16.334)
  ALP : Change at EOS: number analyzed (Participants) | 0 | 13
  ALP : Change at EOS |  | 59.12 (20.822)
  Osteocalcin: Change at Week 8: number analyzed (Participants) | 16 | 0
  Osteocalcin: Change at Week 8 | 8.2 (20.24) |
  Osteocalcin: Change at Week 16: number analyzed (Participants) | 0 | 15
  Osteocalcin: Change at Week 16 |  | 10.3 (21.57)
  Osteocalcin: Change at EOS: number analyzed (Participants) | 0 | 13
  Osteocalcin: Change at EOS |  | 94.0 (32.60)
  Sclerostin: Change at Week 8: number analyzed (Participants) | 12 | 0
  Sclerostin: Change at Week 8 | 0.146 (0.1380) |
  Sclerostin: Change at Week 16: number analyzed (Participants) | 0 | 13
  Sclerostin: Change at Week 16 |  | -0.062 (0.0946)
  Sclerostin: Change at EOS: number analyzed (Participants) | 0 | 11
  Sclerostin: Change at EOS |  | -0.051 (0.1037)

13. Secondary Outcome: Change From Baseline in Biochemical Bone Markers for Tartrate-Resistant Acid Phosphatase (TRAP)
Description: Change from baseline in bone turnover markers for, tartrate-resistant acid phosphatase (TRAP) was reported for combined Part 2 and 3. End of the study was defined as the completion if the participants benefited from and desired to continue dosing with lanthanum. Here, number of participants analyzed refers to the number of participants evaluable for this outcome at specified time point. Data was analyzed and presented as per the intervention received in this study related to this outcome and not analyzed based on each part of the study.
Time Frame: Baseline, Week 8, Week 16 and EOS (up to 42 weeks)
Population: as for outcome 6
Measure: Mean (Standard Error); unit: unit per liter (U/L)
Arm/Group | Part 2: Calcium Carbonate | Part 2 + Part 3: Lanthanum Carbonate
Number analyzed (Participants) | 17 | 17
unit per liter (U/L)
  Change at Week 8: number analyzed (Participants) | 16 | 0
  Change at Week 8 | -1.71 (1.141) |
  Change at Week 16: number analyzed (Participants) | 0 | 15
  Change at Week 16 |  | 1.95 (1.173)
  Change at EOS: number analyzed (Participants) | 0 | 13
  Change at EOS |  | 4.65 (1.934)

14. Secondary Outcome: Change From Baseline in Biochemical Bone Markers for Fibroblast Growth Factor 23 (FGF-23)
Description: Change from baseline in bone turnover markers including fibroblast growth factor 23 (FGF-23) was reported for combined Part 2 and 3. End of the study was defined as the completion if the participants benefited from and desired to continue dosing with lanthanum. Here, number of participants analyzed refers to the number of participants evaluable for this outcome at specified time point. Data was analyzed and presented as per the intervention received in this study related to this outcome and not analyzed based on each part of the study.
Time Frame: Baseline, Week 8, Week 16 and EOS (up to 42 weeks)
Population: as for outcome 6
Measure: Mean (Standard Error); unit: relative unit per milliliter (RU/ml)
Arm/Group | Part 2: Calcium Carbonate | Part 2 + Part 3: Lanthanum Carbonate
Number analyzed (Participants) | 17 | 17
relative unit per milliliter (RU/ml)
  Change at Week 8: number analyzed (Participants) | 16 | 0
  Change at Week 8 | 5130.3 (5232.21) |
  Change at Week 16: number analyzed (Participants) | 0 | 15
  Change at Week 16 |  | -8162.4 (5274.60)
  Change at EOS: number analyzed (Participants) | 0 | 13
  Change at EOS |  | -251.1 (1736.51)

15. Secondary Outcome: Change From Baseline in Biochemical Bone Markers for Parathyroid Hormone (PTH)
Description: Change from baseline in bone turnover markers for parathyroid hormone was reported for combined Part 2 and 3. End of the study is the completion if the participants benefited from and desired to continue dosing with lanthanum. Here, number of participants analyzed refers to the number of participants evaluable for this outcome at specified time point. Data was analyzed and presented as per the intervention received in this study related to this outcome and not analyzed based on each part of the study.
Time Frame: Baseline, Week 8, Week 16 and EOS (up to 42 weeks)
Population: as for outcome 6
Measure: Mean (Standard Error); unit: picomole per litre (pmol/L)
Arm/Group | Part 2: Calcium Carbonate | Part 2 + Part 3: Lanthanum Carbonate
Number analyzed (Participants) | 17 | 17
picomole per litre (pmol/L)
  Change at Week 8: number analyzed (Participants) | 16 | 0
  Change at Week 8 | -7.132 (9.7669) |
  Change at Week 16: number analyzed (Participants) | 0 | 15
  Change at Week 16 |  | 16.273 (12.5441)
  Change at EOS: number analyzed (Participants) | 0 | 13
  Change at EOS |  | 59.801 (16.3097)

16. Secondary Outcome: Change From Baseline in Biochemical Bone Markers for Fetuin-A
Description: Change from baseline in bone turnover markers for fetuin-A was reported for combined Part 2 and 3. End of the study is the completion if the participants has benefited from and desires to continue dosing with lanthanum. Here, number of participants analyzed refers to the number of participants evaluable for this outcome at specified time point. Data was analyzed and presented as per the intervention received in this study related to this outcome and not analyzed based on each part of the study.
Time Frame: Baseline, Week 8, Week 16 and EOS (up to 42 weeks)
Population: as for outcome 6
Measure: Mean (Standard Error); unit: gram per liter (g/L)
Arm/Group | Part 2: Calcium Carbonate | Part 2 + Part 3: Lanthanum Carbonate
Number analyzed (Participants) | 17 | 17
gram per liter (g/L)
  Changed at Week 8: number analyzed (Participants) | 12 | 0
  Changed at Week 8 | -0.006 (0.0301) |
  Change at Week 16: number analyzed (Participants) | 0 | 13
  Change at Week 16 |  | 0.037 (0.0360)
  Change at EOS: number analyzed (Participants) | 0 | 11
  Change at EOS |  | 0.039 (0.0273)

17. Secondary Outcome: Change From Baseline in Height
Description: Change from baseline in height for combined Part 2 and Part 3 for each drug at Week 8, 16 and end of study was reported. End of the study was defined as the completion if the participants benefited from and desired to continue dosing with lanthanum. Here, number of participants analyzed refers to the number of participants evaluable for this outcome at specified time point. Data was analyzed and presented as per the intervention received in this study related to this outcome and not analyzed based on each part of the study.
Time Frame: Baseline, Week 8, Week 16, and EOS (up to 42 weeks)
Population: as for outcome 6
Measure: Mean (Standard Error); unit: centimeter (cm)
Arm/Group | Part 2: Calcium Carbonate | Part 2 + Part 3: Lanthanum Carbonate
Number analyzed (Participants) | 17 | 17
centimeter (cm)
  Change at Week 8: number analyzed (Participants) | 17 | 0
  Change at Week 8 | 0.7 (0.39) |
  Change at Week 16: number analyzed (Participants) | 0 | 17
  Change at Week 16 |  | 0.6 (0.25)
  Change at EOS: number analyzed (Participants) | 0 | 13
  Change at EOS |  | 1.3 (0.46)

18. Secondary Outcome: Change From Baseline in Weight
Description: Change from baseline in weight for combined Part 2 and Part 3 for each drug at Week 8, 16 and end of study was reported. End of the study was defined as the completion if the participants benefited from and desired to continue dosing with lanthanum. Here, number of participants analyzed refers to the number of participants evaluable for this outcome at specified time point. Data was analyzed and presented as per the intervention received in this study related to this outcome and not analyzed based on each part of the study.
Time Frame: Baseline, Week 8, Week 16, and EOS (up to 42 weeks)
Population: as for outcome 6
Measure: Mean (Standard Error); unit: kilogram (Kg)
Arm/Group | Part 2: Calcium Carbonate | Part 2 + Part 3: Lanthanum Carbonate
Number analyzed (Participants) | 17 | 17
kilogram (Kg)
  Change at Week 8: number analyzed (Participants) | 17 | 0
  Change at Week 8 | 1.18 (0.524) |
  Change at Week 16: number analyzed (Participants) | 0 | 17
  Change at Week 16 |  | 1.09 (0.358)
  Change at EOS: number analyzed (Participants) | 0 | 13
  Change at EOS |  | 2.86 (0.606)

ADVERSE EVENTS:
Time Frame: From start of study drug administration up to 42 Weeks
Description: SAS1 and SAS2 included all participants who had taken 1 dose of investigational product in Part 1 for SAS 1, Part 2 or 3 for SAS 2 and who had completed at least 1 follow-up safety assessment. Data was presented as per the intervention received in this study and not analyzed based on each part of the study. Lanthanum carbonate data was combined and analysed for part 2 and 3 in the entire study and separately for Part 1.
Groups:
- Part 1: Lanthanum Carbonate: Participants aged 10 to 12 years received 500 mg and greater than (>) 12 years received 1000 mg single dose of lanthanum carbonate oral powder.
Arm/Group | Part 1: Lanthanum Carbonate | Part 2: Calcium Carbonate | Part 2 + Part 3: Lanthanum Carbonate
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/53 | 0/52
Serious Adverse Events (participants affected / at risk) | 0/20 | 9/53 | 19/52
Other Adverse Events (participants affected / at risk) | 2/20 | 10/53 | 20/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: Lanthanum Carbonate (N=20) | Part 2: Calcium Carbonate (N=53) | Part 2 + Part 3: Lanthanum Carbonate (N=52)
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 2 (2) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Device occlusion (General disorders) | 0 (0) | 1 (1) | 1 (1)
Thrombosis in device (General disorders) | 0 (0) | 0 (0) | 1 (1)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Appendicitis perforated (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Catheter site infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (3)
Erysipelas (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Peritonitis (Infections and infestations) | 0 (0) | 0 (0) | 5 (6)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Arteriovenous fistula site haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Graft haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Blood phosphorus (Investigations) | 0 (0) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Hepatitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Fluid overload (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (3)
Metabolic disorder (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: Lanthanum Carbonate (N=20) | Part 2: Calcium Carbonate (N=53) | Part 2 + Part 3: Lanthanum Carbonate (N=52)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 3 (5)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (2) | 5 (6)
Respiratory tract infection (Infections and infestations) | 0 (0) | 3 (4) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 5 (5)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 9 (9) | 5 (9)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 3 (6)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 3 (4) | 6 (9)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Data was analyzed and presented as per the intervention received in this study and not analyzed based on each part of the study. Lanthanum carbonate data was combined and analysed for Part 2 and 3 in the entire study and separately for Part 1.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually

DOCUMENTS (2):
  • Study Protocol (2016-10-18): https://cdn.clinicaltrials.gov/large-docs/79/NCT01696279/Prot_000.pdf
  • Statistical Analysis Plan (2019-02-14): https://cdn.clinicaltrials.gov/large-docs/79/NCT01696279/SAP_001.pdf